CLINICAL TRIAL: NCT04243850
Title: A Single-center, Prospective, Placebo-controlled, Double-blind, Randomized, Cross-over Mechanistic Intervention Study to Investigate the Effect of Empagliflozin on Kidney Function in People With Either Preserved or Impaired Kidney Function With or Without Type 2 Diabetes
Brief Title: REGROUP: Renohemodynamic Effects empaGliflozin in vaRiOUs Populations
Acronym: REGROUP
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, D van Raalte, Principle Investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DC2019REGROUP01
Record Dates: First submitted 2020-01-21; First posted 2020-01-28 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Diabetes Mellitus, Type 2; Chronic Kidney Diseases
Keywords: Sodium Glucose Cotransporter 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: A single-center, prospective, placebo-controlled, double-blind, randomized, cross-over mechanistic intervention study to investigate the effect of empagliflozin on kidney function in people with either preserved or impaired renal function with or without type 2 diabetes
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin (Experimental): Empagliflozine 7 days
  Interventions: Drug: Empagliflozin 10 MG; Drug: Placebo oral tablet; Diagnostic Test: Caffeine
- Placebo (Placebo Comparator): Placebo 7 days
  Interventions: Drug: Empagliflozin 10 MG; Drug: Placebo oral tablet; Diagnostic Test: Caffeine

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Jardiance
Drug: Placebo oral tablet — Placebo
Diagnostic Test: Caffeine — caffeine iv to investigate wheter the changes in renal hemodynamics are adenosine dependent

SUMMARY:
Worldwide, diabetic kidney disease (DKD) is the most common cause of chronic and end stage kidney disease. Large-sized prospective randomized clinical trials indicate that intensified glucose and blood pressure control, the latter especially by using agents that interfere with the renin-angiotensin-aldosterone system (RAS), halts the onset and (particularly) the progression of DKD, in both type 1 Diabetes Mellitus (T1DM) and type 2 Diabetes Mellitus (T2DM) patients. However, despite the wide use of angiotensin-converting enzyme (ACE) inhibitors and angiotensin receptor blockers (ARBs), a considerable amount of patients develop DKD (20-40%), indicating an unmet need for renoprotective therapies as DKD largely causes the increased mortality risk from cardiovascular disease (CVD) in people with diabetes.

Sodium-glucose linked transporters (SGLT-2) inhibitors are a relatively novel glucose-lowering drug for the treatment of T2DM as they lower plasma glucose levels by blocking renal glucose reabsorption. In addition, these agents exert pleiotropic actions beyond glucose control. As such, SGLT-2 inhibitors decrease proximal sodium reabsorption, reduce blood pressure, body weight and uric acid. In large trials and likely through these pleiotropic effects, SGLT2 inhibitors reduce cardiovascular mortality, hospitalization for heart failure and reduce end stage kidney disease. At this point in time, the renoprotective mechanisms involved with SGLT-2 inhibition still remain speculative, though a consistent finding is that SGLT-2 inhibitors reduce estimated eGFR after first dosing, which is reversible after treatment cessation. This "dip" indicates a renal hemodynamic phenomenon reminiscent of the RAS blockers and is thought to reflect a reduction in intraglomerular pressure.

The mechanisms of this observation have only been partially investigated by us and others. From studies in peolpe with T1DM it is hypothesized that SGLT-2 inhibition increases sodium chloride delivery to the macula densa, which in turn augments the afferent arteriolar resistances, known as tubuloglomerular feedback (TGF), consequently reducing glomerular (hyper)filtration and hydrostatic pressure. Recently a trial has been conducted in humans with T2DM to investigate if this also holds true in these patients. Suprisingly, this study showed that the renohemodynamic actions of SGLT-2 inhibition in T2DM are not due to afferent vasoconstriction but rather efferent vasodilation [van Bommel/van Raalte Kidney International 2019 in press]. The investigators realized that the SGLT-2 associated dip in eGFR remains insufficient understood. The increase in sodium excretion following SGLT-2 inhibition peaks at day 2-3 after which it normalizes. It is unknown whether this drop in eGFR is related to this peak in sodium excretion, as the drop remains after normalization of sodium excretion. Therefore it might be possible that glucosuria, by inducing osmotic diuresis, is the main driver of the reduction in intraglomerular pressure more than sodium, since SGLT-2 inhibitors cause persisting glucosuria.

Furthermore, it is known that SGLT-2 induced glucosuria and possibly sodium excretion is dependent of renal function and HbA1c and consequently is diminished in people with CKD or without T2DM. However, the renoprotective effects in T2DM are also observed in patients with impaired kidney function and seem statistically independent of glucose levels. Until now it has not been investigated whether or not the SGLT-2 induced eGFR alterations occur in people with CKD with or without T2DM. It is clinically relevant to understand the renal hemodynamics of SGLT-2 inhibitors in these populations since then it is possible to interpret the results from the ongoing trials in people with CKD without T2DM, such as EMPA-KIDNEY and DAPA-CKD.

Recently, potential mediators of renal arterole tone, such as adenosine, have been measured to gain more insight into mechanisms of SGLT-2 inhibitor-induced changes in renal hemodynamics. Adenosine is known to augment preglomerular arteriolar resistance. Adenosine was significantly increased after SGLT-2 inhibition, as was also observed in patients with type 1 diabetes. However, it can also induce postglomerular vasodilation via A2aR activation in the presence of RAS blockade. One study in T1DM rats has shown that increased adenosine generation by the macula densa in response to SGLT-2 inhibition suppresses hyperfiltration, as the improvements in preglomerular arteriolar resistance were abolished after adenosine antagonist administration. To date, this has not been investigated in T2DM humans. Therefore, this trial will assess TGF responses with and without adenosine blockade by caffeine.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian*
* Both genders (females must be post-menopausal; no menses >1 year; in case of doubt, Follicle-Stimulating Hormone (FSH) will be determined with cut-off defined as >31 U/L)
* Age: 45 - 80 years
* BMI: >25 kg/m2
* For with people with diabetes - a diagnosis of T2DM with glycosylated haemoglobin (HbA1c) ≥6.5% (≥48 mmol/mol) and <10.5% (<91 mmol/mol); and eGFR (CKD-EPI) between ≥25 and ≤50 mL/min/1.73m2 or >75 mL/min/1.73m2 at the Screening Visit (Visit 1).
* In the normoglycemic, hypertensive, individuals: HbA1c <6.5% (<48 mmol/mol) and an eGFR (CKD-EPI) between ≥25 and ≤50 mL/min/1.73m2 at the Screening Visit (Visit 1).
* In the diabetic arm: people with an eGFR >75 ml/min/1.73m2 should be treated with a stable dose of metformin and/or SU, people with an eGFR between ≥25 and ≤50 mL/min/1.73m2 should be treated with a stable dose of metformin, SU and/or insulin therapy for at least 3 months prior to inclusion
* Patient specific antihypertensive dose of an angiotensin receptor blocker (ARB) (as per Investigator's judgement) for at least 4 weeks prior to Visit 2 (Day 3).
* Written informed consent

Exclusion Criteria:

* History of unstable or rapidly progressing renal disease
* Macroalbuminuria; defined as ACR of 300mg/g.
* Diagnosis of polycystic kidney disease.
* Post renal transplant
* History of or current lupus nephritis.
* Abnormal vital signs, after 10 minutes supine rest, definas as any of the following (Visit 1):

  * Systolic blood pressure above 180 mmHg
  * Diastolic blood pressure above 110 mmHg
* Current/chronic use of the following medication: SGLT2 inhibitors,TZD, GLP-1RA, DPP-4 inhibitors, , antimicrobial agents or chemotherapeutics.
* Volume depleted patients. Patients at risk for volume depletion due to co-existing conditions or concomitant medications, such as loop diuretics should have careful monitoring of their volume status.
* Chronic use of non-steroidal anti-inflammatory drugs (NSAIDs) will not be allowed, unless used as incidental medication (1-2 tablets) for non-chronic indications (i.e. sports injury, head-ache or back ache). However, no such drug can be taken within a time-frame of 2 weeks prior to renal-testing
* History of diabetic ketoacidosis (DKA) requiring medical intervention (e.g. emergency room visit and/or hospitalization) within 1 month prior to the Screening visit.
* Current urinary tract infection and active nephritis
* Recent (<3 months) history of cardiovascular disease, including:

  * Acute coronary syndrome
  * Chronic heart failure (New York Heart Association grade II-IV)
  * Stroke or transient ischemic neurologic disorder
* Complaints compatible with neurogenic bladder and/or incomplete bladder emptying (as determined by ultrasonic bladder scan)
* Severe hepatic insufficiency and/or significant abnormal liver function defined as aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >3x ULN
* History of or actual malignancy (except basal cell carcinoma)
* History of or actual severe mental disease
* Substance abuse (alcohol: defined as >4 units/day)
* Allergy to any of the agents used in the study

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
measured glomerulair filtration rate (mGFR) | 7 days
  using iohexol

SECONDARY OUTCOMES:
effective renal plasma flow | 7 days
  as part of renal hemodynamics
renal vascular resistance | 7 days
  as part of renal hemodynamics
Caffeine-induced changes in renal hemodynamics | 7 days
  to investigate whether the observed changes are adenosine dependent
proximal sodium excretion | 7 days
  using fractional excretion of lithium as a surrogate of proximal sodium handling

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818